CLINICAL TRIAL: NCT00495495
Title: A Multi-Center Study to Evaluate the Safety and Efficacy of the Use of Ozone for the Management of Fissure Caries
Brief Title: Healozone Study to Evaluate the Safety and Efficacy of the Use of Ozone for Management of Dental Caries
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Tufts University School of Dental Medicine (Other); State University of New York at Buffalo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 07-D-187; IDE G50008; Clinical Trials. gov (Registry Identifier: ClinicalTrials.gov protocol registration system)
Record Dates: First submitted 2007-07-01; First posted 2007-07-03 (Estimated); Results first posted 2010-12-23 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ozone treatment (Experimental): Ozone treatment of randomly selected study tooth for 60 seconds
  Interventions: Device: Ozone treatment
- Placebo, no ozone (Placebo Comparator): Placebo treatment (no ozone) of randomly selected study tooth for 60 seconds.
  Interventions: Device: Placebo treatment

INTERVENTIONS:
Device: Ozone treatment — Ozone treatment applied to randomly selected tooth for a period of 60 seconds at Baseline, Three, Six and Nine-Month visits.
  Other Names: HealOzone unit
  Arms: Ozone treatment
Device: Placebo treatment — Placebo treatment applied to randomly selected tooth for a period of 60 seconds at Baseline, Three-, Six- and Nine-Month visits.
  Arms: Placebo, no ozone

SUMMARY:
Caries means demineralization with the formation of cavities and pulp symptoms and necrosis as an end result. The acids in the mouth are mainly produced by oral bacteria like Streptococcus mutans from bacterial biofilms adhering to the tooth. Ozone has been shown to have a very strong bactericidal effect on bacteria causing dental caries. Baysan et al reported that there was a statistically significant reduction of streptococci in root caries lesions and saliva samples after ozone application. The positive clinical effect of ozone with respect to arresting caries progression and the remineralization of caries has been shown in vitro and in vivo. In an in vivo study, Baysan and Lynch found that the application of ozone resulted in a significant reduction of bacterial contamination as well as a reduction in size and severity of root caries lesions. In a subsequent study, Baysan and Lynch reported that the severity of root caries lesions was significantly reduced after ozone application as measured by electrical conductance and laser fluorescence. In several studies, the caries reducing effect of ozone was measured with biochemical methods in root surface caries lesions, the biofilm and saliva after ozone application. See Citation section for references.

The objectives of this multi-center clinical study were to determine: (1) the effectiveness of the HealOzone in stopping the progression of fissure caries; and (2) the oral soft tissue safety of the ozone system.

DETAILED DESCRIPTION:
The proposed study was designed as a twelve-month, multi-center, double-blind, randomized controlled clinical study involving 394 subjects with 788 lesions. There were three sites participating in this trial: Indiana University School of Dentistry (lead site), Tufts University School of Dental Medicine, and SUNY School of Dental Medicine. Each site submitted a version of the protocol to their respective Institutional Review Board ("IRB") that incorporated the specific institutional and state guidelines and regulations applicable to that site.

The two treatment regimens were: (a) placebo treatment and (b) experimental ozone treatment. Selected subjects had to have at least two teeth with similar stages of early active fissure caries. The selection of the study teeth was determined by a review of the visual examination, including the ICDAS severity score and the caries lesion activity score, conducted at the screening visit, in conjunction with the bitewing radiographs. The decision whether a tooth was to be treated with ozone or receive placebo treatment was made randomly.

All clinical personnel involved in the clinical examinations and treatment application were trained at the primary site prior to the initiation of the trial both in the use of the device, and in how to identify the signs and symptoms of ozone toxicity and in how to provide the appropriate medical response should any of these signs or symptoms be observed.

All qualified subjects received the following:

1. Professional dental cleaning and scaling at the Screening Visit (or separate visit prior to baseline visit and after completing the study at 12 months.
2. Diagnostic procedures:

   1. Clinical visual examination (utilizing the International Caries Detection and Assessment System [ICDAS] severity scoring)
   2. Clinical visual/tactile assessment of caries lesion activity
   3. Bitewing x-rays
   4. Laser fluorescence measurement (utilizing the DIAGNOdent, KaVo)
3. Treatment Regimen:

Using a split-mouth design, the assigned investigational treatment regimen was administered on the two selected study teeth at the baseline, and at the three-, six- and nine-month appointments.

After three, six, nine and twelve months, the diagnostic procedures were repeated with the exception of bitewing x-rays, which were only repeated at the twelve-month exam (unless the examining dentist determined that x-rays also were needed at the six- or nine-month visit to confirm whether dentinal caries were present). In addition, optional digital photographs were taken at the Boston site of selected study teeth to document clinical changes over the study period.

If a selected study tooth progressed from an initial caries lesion to a more advanced lesion, which in the judgment of the examining dentist required restorative intervention, the tooth was restored at no cost to the subject and the lesion was recorded as 'progression from baseline' at any remaining examinations. The subject was eligible to remain in the study.

Subjects received a thorough dental cleaning and scaling and topical fluoride treatment at the conclusion of the twelve-month examination.

The primary efficacy parameter will be the ICDAS severity value. The severity criteria used in the ICDAS diagnostic system are as follows:

0 = Sound tooth surface.

1. = First visual change in enamel.
2. = Distinct visual change in enamel.
3. = Localized enamel breakdown due to caries with no visible dentin.
4. = Underlying dark shadow from dentin, with or without localized enamel breakdown.
5. = Distinct cavity with visible dentin.
6. = Extensive distinct cavity with visible dentin.

The secondary efficacy parameters will be measured by:

Caries Lesion Activity score:

1. = Inactive - surface of enamel appears whitish, brownish or black. Enamel may be shiny and feels hard and smooth when the tip of the probe is moved gently across the surface.
2. = Active lesion - surface of enamel appears whitish/yellowish opaque with loss of luster. The surface feels rough when the tip of the probe is moved gently across the surface.

Radiographic Changes:

The occlusal surface of study teeth will be evaluated using the following scale:

Lesion presence: yes /no

Lesion depth:

E1 = outer half of enamel E2 = inner half of enamel D1 = outer third of dentin D2 = middle third of dentin D3 = inner third of dentin or greater/pulpal exposure

Laser fluorescence measurement:

DIAGNOdent reading using a scale from 00 to 99, with 00 indicating no caries activity and 99 indicating a high level of activity.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for study participation, subjects had to:

1. provide written informed consent, HIPAA authorization and medical history information prior to their participation; 2. be between the ages of 10 and 40 years of age; 3. if female and of childbearing potential, agree to:

* a urine pregnancy test, which must be negative;
* use one form of medically accepted contraceptive measures which include oral contraceptives, condom, or diaphragm with spermicide, Intra Uterine Device (IUD), Depo-Provera, Norplant during the study and for at least 30 days after the last treatment. (Females who are post menopausal, i.e. amenorrhea for the previous 12 months, or surgically sterile may be included.) 4. be in good general health as evidenced by a review of the medical history; 5. have good oral health; 6. agree to comply with all subjects' responsibilities as stated in the protocol (e.g. attendance at appointments, turning off of cell phone during appointment, etc.); and 7. have two posterior (molar or premolar) teeth with active fissure caries as defined by ICDAS severity score between 1 and 4, a caries lesion activity score of 2, and with radiographic evidence indicating that there is no extension past the dentinal enamel junction. Lesions within the same subject ideally should have the same ICDAS criterion; however, the following deviations will be acceptable - teeth with ICDAS criterion 1 paired with a 2, and a 3 paired with a 4.

Exclusion Criteria:

Any of the following excluded subjects from participating:

1. a medical condition that requires antibiotic therapy prior to dental work;
2. any medical condition that could be expected to interfere with the subject's safety, such as a pacemaker or similar powered implant;
3. selected study teeth with occlusal restorations, sealants, carious lesions extending into dentin, hypomineralization or fluorosis;
4. generalized severe gingivitis or gross unrestored caries;
5. orthodontic appliances that interfere with access to selected study teeth;
6. pregnant or nursing.

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 394 (Actual)
Dates: Start 2007-02; Primary Completion 2009-05 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Domenick T Zero, DDS MS, Principal Investigator — Indiana University; Athena Papas, DMD, PhD, Principal Investigator — Tufts University School of Dental Medicine; Sebastian Ciancio, DDS, PhD, Principal Investigator — SUNY School of Dental Medicine
Locations (3):
- United States (3):
  - Indiana University School of Dentistry, Indianapolis, Indiana
  - Tufts University School of Dental Medicine, Boston, Massachusetts
  - State University of New York at Buffalo, School of Dental Medicine, Buffalo, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Ozone Treatment and Placebo Treatment: 60-second Ozone device treatment compared to 60-second Placebo device treatment. Study utilized split-mouth design. The paired treatment assignment for the two teeth within each subject was performed according to a randomization table provided by the Biometrician. Randomization of teeth to Ozone treatment or Placebo treatment was stratifed according to tooth similarity.
Period: Overall Study
Arm/Group | Ozone Treatment and Placebo Treatment
Started | 394
Completed | 295
Not Completed | 99
Not completed — Protocol Violation | 99

BASELINE CHARACTERISTICS:
Groups:
- Ozone Treatment/Placebo Treatment: Study utilized split-mouth design. Each participant had two teeth selected at the start of the study. Each participant was then randomized to receive Ozone treatment on a randomly selected study tooth for 60 seconds and Placebo treatment on a randomly selected study tooth for 60 seconds.
Arm/Group | Ozone Treatment/Placebo Treatment
Number analyzed (Participants) | 394
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 102
  Between 18 and 65 years | 292
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.9 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202
  Male | 192
Region of Enrollment [Number; unit: participants]
  United States | 394

OUTCOME MEASURES:

1. Primary Outcome: ICDAS Severity Value
Description: Clinically significant changes indicating caries progression are defined as changes in ICDAS severity values from 1 or 2 to a 3 or higher, or from a 3 or 4 to a 5 or higher. The severity criteria are as follows:
  0 = Sound tooth surface.
  1. = First visual change in enamel.
  2. = Distinct visual change in enamel.
  3. = Localized enamel breakdown due to caries with no visible dentin.
  4. = Underlying dark shadow from dentin, with or without localized enamel breakdown.
  5. = Distinct cavity with visible dentin.
  6. = Extensive distinct cavity with visible dentin.
Time Frame: Baseline and One Year
Population: The study utilized a split-mouth design. The results posted are for the Per Protocol dataset. Subjects who completed all four treatment/examination visits as well as final examination visit without major protocol violations were included in this dataset.
Measure: Number; unit: teeth
Units Other Than Participants: teeth
Groups:
- Ozone Treatment: As part of the split-mouth design, subjects were randomized to receive Ozone treatment on a randomly selected study tooth for 60 seconds.
- Placebo Treatment: As part of the split-mouth design, subjects were randomized to receive placebo treatment on a randomly selected study tooth for 60 seconds.
Arm/Group | Ozone Treatment | Placebo Treatment
Number analyzed (Participants) | 295 | 295
Number analyzed (teeth) | 295 | 295
teeth
  Number of Teeth with Caries Progression | 17 | 22
  Number of Teeth with No Caries Progression | 278 | 273
Statistical Analysis 1: Comparison: Ozone Treatment; Null hypothesis: there is no difference between the HealOzone and Placebo devices in the proportion of teeth with lesion progression after 1 year. Power calculation: the study was sized to have 90% power to detect a 15% difference between treatments in the percentage of teeth with lesion progression at one year (i.e., assuming 45% for the lesions treated with the Placebo device and 30% for the lesions treated with the HealOzone device) with a sample size of 258 subjects completing the study; Test type: Superiority or Other; p = 0.1126, McNemar; Risk Difference (RD) = .02

2. Secondary Outcome: Change in Caries Lesion Activity
Description: Change in caries lesion activity at One Year. All teeth were considered Active at Baseline
  Caries Lesion Activity score:
  1. = Inactive - surface of enamel appears whitish, brownish or black. Enamel may be shiny and feels hard and smooth when the tip of the probe is moved gently across the surface.
  2. = Active lesion - surface of enamel appears whitish/yellowish opaque with loss of luster. The surface feels rough when the tip of the probe is moved gently across the surface.
Time Frame: Baseline and one year
Population: Analyses were based on per protocol subjects, defined as all randomized subjects with no major protocol violations.
  Clinically significant changes for Activity Scores were indicated by a change in caries activity status from active to inactive. It should be noted that all teeth were considered active at baseline.
Measure: Number; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Ozone Treatment | Placebo Treatment
Number analyzed (Participants) | 295 | 295
Number analyzed (teeth) | 295 | 295
teeth
  Number of Active Caries lesions | 189 | 164
  Number of Non- Active Caries Lesions | 106 | 131
Statistical Analysis 1: Comparison: Ozone Treatment vs Placebo Treatment; Test type: Superiority or Other; p = .9777, McNemar; Risk Difference (RD) = .08

3. Secondary Outcome: Progression of Radiographic Scores at 12 Months
Description: Clinically significant changes for Bitewing x-rays indicating caries progression would be changes in x-ray criterion for lesion presence from "no" to "yes" or for lesion depth to a D1 or higher. The occlusal surface of study teeth will be evaluated using the following scale:
  Lesion presence: yes /no
  Lesion depth:
  E1 = outer half of enamel E2 = inner half of enamel D1 = outer third of dentin D2 = middle third of dentin D3 = inner third of dentin or greater/pulpal exposure
Time Frame: one year
Population: Analyses were based on per protocol subjects, defined as all randomized subjects with no major protocol violations (subjects who completed all four treatment/examination visit at Baseline, 3-, 6-, 9-month as well as Final examination at 12-month.
Measure: Number; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Ozone Treatment | Placebo Treatment
Number analyzed (Participants) | 295 | 295
Number analyzed (teeth) | 295 | 295
teeth
  Number of Teeth with Progression | 6 | 12
  Number of Teeth with No Progression | 220 | 214
Statistical Analysis 1: Comparison: Ozone Treatment vs Placebo Treatment; Test type: Superiority or Other; p = .0416, McNemar

4. Secondary Outcome: Laser Fluorescence Progression-12 Month (Increase From <=20 to >=30)
Description: The change in DIAGNOdent measurements between baseline and twelve-month visits was used as an additional secondary endpoint. Clinically significant changes for DIAGNOdent indicating caries progression would be an increase in DIAGNOdent reading of 10 or more units or an increase in DIAGNOdent reading from below 20 to above 30 units. DIAGNOdent reading using a scale from 00 to 99, with 00 indicating no caries activity and 99 indicating a high level of activity.
Time Frame: one year
Population: as for outcome 3
Measure: Number; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Ozone Treatment | Placebo Treatment
Number analyzed (Participants) | 293 | 293
Number analyzed (teeth) | 293 | 293
teeth
  Number of Teeth with Progression | 16 | 14
  Number of Teeth with No Progression | 277 | 279
Statistical Analysis 1: Comparison: Ozone Treatment vs Placebo Treatment; Test type: Superiority or Other; p = 0.6585, McNemar; Risk Difference (RD) = .01

5. Secondary Outcome: Laser Fluorescence Progression-12 Month (Increase at Least 10)
Description: The change in DIAGNOdent measurements between baseline and twelve-month visits was used as an additional secondary endpoint. Clinically significant changes for DIAGNOdent indicating caries progression would be an increase in DIAGNOdent reading of 10 or more units. DIAGNOdent reading using a scale from 00 to 99, with 00 indicating no caries activity and 99 indicating a high level of activity.
Time Frame: one year
Population: Analyses were based on per protocol subjects, defined as all randomized subjects with no major protocol violations.
Measure: Number; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Ozone Treatment | Placebo Treatment
Number analyzed (Participants) | 293 | 293
Number analyzed (teeth) | 293 | 293
teeth
  Number of Teeth with Progression | 58 | 52
  Number of Teeth with No Progression | 235 | 241
Statistical Analysis 1: Comparison: Ozone Treatment vs Placebo Treatment; Test type: Superiority or Other; p = .7666, McNemar; Risk Difference (RD) = .02

ADVERSE EVENTS:
Time Frame: The adverse events were collected during the one-year period of the trial.
Groups:
- Ozone Treatment and Placebo Treatment: Study utilized split-mouth design. Each participant had two teeth selected at the start of the study. Each participant was then randominzed to receive Ozone treatment on a randomly selected study tooth for 60 seconds and Placebo treatment on a randomly selected study tooth for 60 seconds.
Arm/Group | Ozone Treatment and Placebo Treatment
Serious Adverse Events (participants affected / at risk) | 5/394
Other Adverse Events (participants affected / at risk) | 0/394
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ozone Treatment and Placebo Treatment (N=394)
Appendicitis (General disorders) | 1 (1) — Not related to ozone device
Surgery ovarian cyst removal (Reproductive system and breast disorders) | 1 (1) — Not related to ozone device
surgery breast reduction (Reproductive system and breast disorders) | 1 (1) — Not related to ozone device
Broken left leg (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to ozone device
Broken left knee (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to ozone device

LIMITATIONS AND CAVEATS:
Study length may have been too brief to permit progression of early stage caries; Low caries increment in study population; Difficult to establish that lesions were truly active at baseline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No